CLINICAL TRIAL: NCT04391062
Title: A Multi-center Phase II Study With Light Dose Escalation During Intraoperative Photodynamic Therapy of Glioblastoma
Brief Title: Dose Finding for Intraoperative Photodynamic Therapy of Glioblastoma
Acronym: DOSINDYGO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government); Hemerion Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2018_58; 2019-004796-40 (EudraCT Number); 2019-A03157-50 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2020-05-12; First posted 2020-05-18 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Glioblastoma
Keywords: Surgical indication of glioblastoma; Glioblastoma; Photodynamic Therapy; Neurosurgery; Oncology; 5-aminolevulinic Acid
MeSH Terms: conditions — Glioblastoma; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- intraoperative PDT 400J/cm² (Experimental)
  Interventions: Drug: Gliolan; Device: Intraoperative PDT
- intraoperative PDT 600J/cm² (Experimental)
  Interventions: Drug: Gliolan; Device: Intraoperative PDT
- intraoperative PDT 800J/cm² (Experimental)
  Interventions: Drug: Gliolan; Device: Intraoperative PDT

INTERVENTIONS:
Drug: Gliolan — patient will receive 5-ALA 4 to 6 hours before surgery
Device: Intraoperative PDT — The protocol requires the realization of specific procedures in addition to the usual care.
  The intra-operative photodynamic therapy ("intraoperative PDT") added to surgery for glioblastoma excision. The patient will receive 5-ALA ( 5-aminolevulinic acid hydrochloride),GLIOLAN drinkable 6h before surgery + lighting of the tumor bed by a red light source (laser with different J/cm²) at the end of resection (Prolonged surgery of 45 minutes).

SUMMARY:
The phase II study evaluate a light dose escalation in a classical intraoperative PDT regimen mediated by 5-ALA-PpIX, in glioblastoma patients with access to full surgical removal of the contrast enhancement. This treatment will be performed in addition to the current reference treatment of glioblastoma: maximum removal surgery followed by radiochemotherapy according to the Stupp protocol.

ELIGIBILITY:
Inclusion Criteria:

* General status (WHO) Karnofsky Performance Status ≥60
* Presumptive glioblastoma according to radiological criteria,
* Surgical indication decided in Multidisciplinary consultation meeting (RCP) of neuro oncology,
* Decision to treat the patient as part of the Clinical trial achieved in neuro-oncology RCP ("Multidisciplinary consultation meeting")
* Patient operable on the basis of absence of cardiopulmonary disease history; a complete medical check-up sufficient to insure a post-operative state with normal daily life
* Clinical neuro-oncological monitoring and long-term MRI/ TEP 11C MET scheduled at the hospital centers
* Patient able to understand and sign voluntarily Informed consent
* Patient able to adhere to the visit's calendar of the study and other imperatives of the protocol
* Women of child-bearing potential should benefit of an effective contraception
* For patients receiving hepatotoxic therapy in the long term, this treatment must be suspended during the 24h after taking 5-ALA

Exclusion Criteria:

* Contraindications to 5-ALA (Gliolan®) and to intra-operative PhotoDynamic Therapy "intraoperative PDT":
* Contraindications to 5-ALA

  * Porphyria
  * Taking photosensitizer treatment
  * Severe renal or hepatic impairment
  * Bilirubin> 1.5 x maximum level, Alkaline Phosphatases and transaminases (ASAT)> 2.5 x Maximum. rates
  * Creatinine clearance <30 mL / min;
  * Non-compliance with the rules of prevention of the transient risk of cutaneous photosensitization
* Contraindications to surgery
* Contraindications to magnetic resonance imaging (MRI/TEP 11C MET
* Treatment with an experimental drug within 30 Days prior to the start of the study
* Clinical follow-up impossible to perform for psychological, familial, social or geographical reasons,
* Legal incapacity (persons deprived of their liberty or Guardianship or guardianship),
* Pregnant or nursing women
* Refusal to participate or sign the consent of the study
* Soy allergy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2021-09-28 (Actual); Primary Completion 2024-03-25 (Actual); Study Completion 2024-03-25 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose-Light Level (MTDL) defined as the light dose associated with an acceptable dose-limiting toxicity level (TDL) | 4 weeks (+/-3 days) post-PDT.
  Dose level above which TDL is observed in more than 33% (i.e., d̀-> 2 of 6) of subjects in an arm

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | From the Date of diagnosis of glioblastoma until the date of Relapse, an average 18 months
  Number of patients without relapse within 25 mm of surgical site defined according to International RANO criteria
Global Progression Free Survival (PFS) | From the Date of diagnosis of glioblastoma until the date of Relapse, an average 18 months
  Median of progression-free survival time determined according to international RANO criteria
Overall Survival (OS) | From the Date of diagnosis of glioblastoma until the death, an average 18 months
  Median of OS determined according to international RANO criteria
Response to treatment | every 3 months between the Date of intraoperative PDT until relapse/death, an average 18 months
  Evaluated by MRI/ TEP 11C-MET every 3 months
Incidence of "intraoperative PDT" treatment-emergent Adverse Events | From the beginning of treatment with intraoperative PDT up to relapsing/death, an average 18 months
  Collection of all Adverse events (AEs and SAEs) (according to NCI-CTCE V5.0) and reviewing by an Independent Safety Monitoring Board
Quality of Life Questionnaire -C30 ( QLQ-C30 | Every 3 months from the signature of Consent form until relapse/death, an average 18 months
  The QLQ-C30 is composed of both multi-item scales and single-item measures. These include five functional scales, three symptom scales, a global health status / QoL scale, and six single items
Quality of Life Questionnaire - Brain Cancer Module (QLQ-BN20) | Every 3 months from the signature of Consent form until relapse/death, an average 18 months
  Measuring the health-related quality of life in patients with brain cancer

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Reyns, MD,PhD, Principal Investigator — University Hospital, Lille
Locations (2):
- Hôpital Erasme, Clinique Universitaire de Bruxelles, Brussels, Belgium
- Hopital Roger Salengro, CHU Lille, Lille, France